CLINICAL TRIAL: NCT02612896
Title: Taenia Solium Elimination Versus Control: What is the Best Way Forward for Sub-Saharan Africa?
Acronym: CYSTISTOP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Tropical Medicine, Belgium (Other)
Collaborators: University of Zambia (Other); Ministry of Health, Zambia (Other Government); Université Catholique de Louvain (Other); University Ghent (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CYSTISTOP_2.2_07012016
Record Dates: First submitted 2015-11-17; First posted 2015-11-24 (Estimated); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Taenia Solium Infection
Keywords: Taenia solium; control; elimination; One Health
MeSH Terms: conditions — Taeniasis | interventions — Mass Drug Administration; Praziquantel; Educational Status

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Elimination arm (Experimental): Both human and porcine interventions at four-monthly intervals in the first two study years, for a total of six iterations (only human interventions will be detailed here):
  Human: Mass drug administration, praziquantel 10mg/kg, according to the list of WHO recommended anthelmintic drugs for use in preventive chemotherapy for taeniasis. And Health Education
  Interventions: Drug: Mass drug administration, praziquantel 10mg/kg; Behavioral: Health education
- Control intervention arm (Experimental): Human: yearly health education, for a total of five iterations. The intervention on the pig host will not be detailed here)
  Interventions: Behavioral: Health education

INTERVENTIONS:
Drug: Mass drug administration, praziquantel 10mg/kg — see previous, in elimination study arm only
  Other Names: praziquantel
  Arms: Elimination arm
Behavioral: Health education — in all study arms, using village meetings, posters, pamphlets.
  Other Names: education

SUMMARY:
Taenia solium taeniosis/cysticercosis is a neglected zoonotic parasitic disease complex with significant economic and public health impacts, occurring primarily in developing countries. Humans are the carriers of the tapeworm (taeniosis); the normal intermediate pig host develops the metacestode larval stage (porcine cysticercosis). However, people can also act as accidental intermediate hosts and develop human cysticercosis or neurocysticercosis (NCC) when the central nervous system is involved.

The scattered efforts of researchers into evaluation of control programmes in Sub-Saharan Africa (SSA) have focussed on single control options. It is becoming clear that these stand-alone options have the potential to reduce the occurrence of the parasite, however either long term or more integrated efforts seem to be required to reach an elimination status.

The objective of the current study is to evaluate the cost-effectiveness/acceptability of elimination (to be achieved on a short term via integrated measures), and control (single measures, with an elimination goal on a longer term) of T. solium in a highly endemic area in SSA.

This intervention study will entail an elimination study arm in which multiple control options are combined (integrated) aiming at the final human host (Mass drug administration (MDA) and health education) and pig intermediate hosts (pig treatment and vaccination). In a second study arm a single control option will be carried out (pig treatment). In both study arms (health) education will be implemented. At baseline and in the final sampling year, prevalence of human taeniosis/cysticercosis and porcine cysticercosis will be determined in all study villages. Active ongoing surveillance and 6 monthly (biannual) human and pig sampling will be conducted in the elimination study arm, as well as two-yearly (biennial) sampling of the pig intermediate host in the control study arm. Additionally, (open ended) questionnaires and focus group discussions will be administered/held to obtain data on the cost of pig keeping, T. solium, the interventions and the perception/acceptability of the proposed control measures to the local communities.

DETAILED DESCRIPTION:
As T. solium is a zoonosis, it's control will be evaluated in a One Health perspective, tackling both the human and pig host. The study will be carried out in the Katete district, in the Eastern Province of Zambia, an area reported to be endemic for T. solium in both pigs and humans. The pig interventions will not be described here, as requested by ClinicalTrials.gov Suitability of communities in the Katete district was assessed during a pilot survey conducted by the proposers (April 2015).

Two communities were selected that fulfilled all of the eligibility criteria. The Nyembe neighbourhood community (1,210 people, 5 villages, 520 pigs), within the Nyembe Rural Health Centre (RHC) catchment was selected for the elimination study arm; and Chimvira neighbourhood community (1,470 people, 11 villages, 827 pigs), in the Mtandaza Rural Health Centre catchment, was selected for the control study arm.

The interventional study will entail a high-input elimination study arm (E), in which multiple control options targeting both the final (human, mass drug administration, health education) and intermediate (pig) hosts (treatment and vaccination), are combined; and a lower-input control study arm (CI), which will use a single control option targeting only the porcine host (treatment).

Teams of suitably qualified and trained human and veterinary medical staff will go from door-to-door to each household in the study communities.

Procedures will include collection of both qualitative and quantitative data from human participants and pigs; subject-related interventions in both human participants and pigs; and laboratory analysis of collected samples.

For the baseline surveys, one randomly-selected consenting adult member and one randomly-selected assenting (and parental consent) child member (above 5 years) from each household will be sampled (serum: diagnosis of human cysticercosis; and stool: diagnosis of taeniasis), whereas for all subsequent surveys in the elimination arm (see protocol for specific time points), all eligible consenting members of the elimination communities will be invited to participate (stool samples: diagnosis of taeniasis). All eligible consenting members from the control arm will be included at the final study sampling (stool: diagnosis of taeniasis and serum: diagnosis of cysticercosis). It is expected that all age, sex and socioeconomic groups will be equally represented.

For the socio-economic questionnaires, 50% of the households will be randomly selected and the head of the household addressed.

The school based questionnaire will be administered to grade 5-6 children attending school in each of the study communities.

For the perception questionnaires: here also 50% of the households will be targeted (random selection), until data saturation has been reached.

For the focus group discussions (FGD): 6 FGD (3 with each time 10 men, 3 with each time 10 women) will be conducted in the elimination study arm, 12 in the control study arm (6 iterations involving 10 men and 6 iterations involving 10 women), at defined time points (table 1), until data saturation has been reached.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to participate in all aspects of the study, including providing blood and stool samples, participating in a questionnaire survey and group discussions, and taking oral anthelmintic tablets (the latter specific for the elimination arm)
* Willing and able to provide informed consent (signature or thumb print with impartial witness; assent for minors with parental consent).
* Living in, attending school in, or regularly visiting the bore holes present in, the study communities
* Aged five years of age or older
* People without epilepsy

Exclusion Criteria:

* Unwilling or unable to participate in some or all aspects of the study, including providing blood and stool samples, participating in a questionnaire survey and group discussions, or taking oral anthelmintic tablets (the latter specific for the elimination arm)

  * Unwilling or unable to provide written (signature or thumb print with impartial witness) informed consent (or assent for minors)
  * Living outside of, and not regularly visiting, or attending school in, the study communities
  * Children aged four years or younger
  * People with epilepsy (identified cases by the Rural Health Centre, questions included in the registration procedure)
  * Seriously ill individuals (people unable to engage in the normal activities of daily living without assistance because of their illnesses)

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2900 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2021-10 (Actual); Study Completion 2022-02 (Actual)

PRIMARY OUTCOMES:
Change in porcine cysticercosis: in this One Health approach, the primary outcome is not a human measure | Elimination arm: day 0, Year 1, Year 2, Year 2.5, Year 3, Year 3.5, Year 4, Year 4.5, Year 5. Control intervention arm: day 0, Year 2, Year 4,Year 5
  serological measurement of porcine cysticercosis (in pigs), antigen ELISA result: ratio

SECONDARY OUTCOMES:
Change in human cysticercosis active infection (serum: ) | in both study arms: day 0, Year 5.
  human cysticercosis: serological diagnosis: B60/B158 Antigen-ELISA (ratio>1 is positive)
Change in human cysticercosis, exposure to infection (serum) | in both study arms: day 0, year 5
  human cysticercosis: serological diagnosis: Enzyme-linked Electroimmunotransfer blot assay (EITB): number of bands: one band is positive
Change in human taeniasis (stool) | in both study arms: day 0, year 5; elimination study arm: Year 1, Year 2, year 2.5, year 3, year 3.5,year 4, year 4.5 and year 5
  human taeniasis: coprological diagnosis: copro- antigen ELISA: Optical Density (OD) values (with all OD's higher then cutoff= positive) ; copro polymerase chain reaction (PCR) followed by restriction fragment length polymorphism (RFLP) if needed: band result leading to pos/neg. An individual is considered 'POSITIVE' if any of the test results is positive.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Dorny, PhD, Study Chair — Institute of Tropical Medicine, Belgium; Emmanuel Bottieau, PhD, MD, Study Chair — Institute of Tropical Medicine, Belgium
Locations (1):
- Nyembe and Mtandaza Rural Health Centre, Katete, Eastern Province, Zambia